CLINICAL TRIAL: NCT02233452
Title: Management of Neuropathic Chronic Pain With Methadone Combined With Ketamine: Randomized, Double Blind, Active-controlled Clinical Trial
Brief Title: Methadone and Ketamine for Neuropathic Pain Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Santa Casa de Misericórdia de Belo Horizonte (Other); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Juliano Ferreira, PhD, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Methadone plus ketamine
Record Dates: First submitted 2014-08-22; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Methadone; Ketamine; Multimodal analgesia
MeSH Terms: conditions — Neuralgia | interventions — Methadone; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methadone (Active Comparator): Group treated with methadone solution.
  Interventions: Drug: Methadone
- Ketamine (Active Comparator): Group treated with ketamine solution
  Interventions: Drug: Ketamine
- Methadone plus ketamine (Active Comparator): Group treated with methadone plus ketamine solution
  Interventions: Drug: Methadone plus Ketamine

INTERVENTIONS:
Drug: Methadone — The solution of methadone was prepared by mixing 10 ml of methadone (10 mg/ml) and 90 ml of saline 0.9% (Baxter, São Paulo, Brazil)
  Other Names: Methadone hydrochloride, Cristália® (São Paulo, Brazil)
  Arms: Methadone
Drug: Ketamine — The solution of ketamine was prepared by mixing 20 ml of S(+)-ketamine hydrochloride (50 mg/ml, Cristália®, São Paulo, Brazil) and 80 ml of saline 0.9% (Baxter, São Paulo, Brazil), obtaining a concentration of 10 mg/ml of ketamine.
  Other Names: S(+)-ketamine hydrochloride, Cristália®, São Paulo, Brazil
  Arms: Ketamine
Drug: Methadone plus Ketamine — the solution of methadone, ketamine was prepared by mixing 10 ml of methadone hydrochloride (10 mg/ml, Cristália®, São Paulo, Brazil), 20 ml of S(+)-ketamine hydrochloride (50 mg/ml, Cristália®, São Paulo, Brazil) and 70 ml of saline 0.9% (Baxter, São Paulo, Brazil), obtaining a concentration of 1 mg/ml of methadone and 10 mg/ml of ketamine.
  Other Names: methadone and S(+)-ketamine, Cristália®, São Paulo, Brazil
  Arms: Methadone plus ketamine

SUMMARY:
Methadone and ketamine are effective for neuropathic pain management. However, the benefits of the association of both drugs are uncertain. Here, the investigators conducted a randomized, double-blind, in parallel, active controlled clinical trial to test the hypothesis that methadone combined ketamine (methadone/ketamine) is more effective than methadone or ketamine alone in reducing neuropathic pain.

DETAILED DESCRIPTION:
Either oral methadone or ketamine have been used in neuropathic pain management, however, the benefits of the association of both drugs are uncertain. Here, we conducted a randomized, double-blind, in parallel, active controlled clinical trial to test the hypothesis that methadone combined ketamine (methadone/ketamine) is more effective than methadone or ketamine alone in reducing neuropathic pain.

Methods: Fourthly two patients with neuropathic pain refractory to conventional therapy were randomly assigned to receive during three months oral methadone (n= 13), ketamine (n=13) or methadone combined with ketamine (n=13). The primary outcome was pain score on visual analogical scale (VAS) assessed on baseline, 8, 15, 30, 60 and 90 days throughout the treatment, and the secondary outcomes were symptoms of neuropathic pain such as allodynia, burning or shooting pain as well the side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients complaining of pain for more than 6 months with neuropathic pain poorly responsive to drugs used to treat neuropathic pain (i.e. opioid, non-opioid, anticonvulsants, antidepressants), who were 22 to 77 years old

Exclusion Criteria:

* patients with a history of severe psychiatric disorder,
* misuse of illegal drugs or
* hepatic disease

Ages: 22 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome was pain intensity as assessed by visual analogical scale (VAS) scores | 90 days

SECONDARY OUTCOMES:
The secondary outcomes were the presence of burning and/or shooting pain, allodynia and side effects. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Juliano Ferreira, PhD, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- University Hospital in Santa Maria, Santa Maria, Rio Grande do Sul, Brazil